CLINICAL TRIAL: NCT01428128
Title: A Phase II Study of Low Dose Arsenic Trioxide in Patients With Malignancies as a Potential Chemotherapy Protector
Brief Title: Low Dose Arsenic Trioxide as a Potential Chemotherapy Protector
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20110177H
Record Dates: First submitted 2011-06-17; First posted 2011-09-02 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer Other Than Leukemia
MeSH Terms: interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arsenic Trioxide (Experimental)
  Interventions: Drug: Arsenic Trioxide

INTERVENTIONS:
Drug: Arsenic Trioxide — IV; 0.005mg/kg. Infusion on Days -3, -2 and -1 of Chemo Cycles 2, 4, and 6 (if more than 4 cycles received).
  Other Names: Brand name: Trisonex

SUMMARY:
Many types of cancer are treated with chemotherapy drugs and/or radiation therapy. These forms of treatment, however, can also damage normal (non-cancer) cells and cause a variety of side effects. There are many side effects of chemotherapy. A few examples are: lowered red blood cell counts (anemia) which can lead to tiredness, weakness or shortness of breath; lowered white cell counts (white blood cells which help the body to fight infection); low platelet counts (platelets help blood to clot); nausea and vomiting; diarrhea; lip and mouth sores and hair loss. These side effects can range from mild to severe. P53 is a protein in the body that regulates the cell cycle. If a cell becomes damaged from chemotherapy or radiation treatment, the p53 protein becomes activated. This activation can cause the cell to die and is involved in causing side effects from chemotherapy or radiation therapy.

Arsenic trioxide is a drug that is currently approved by the FDA (Food and Drug Administration) for the treatment of acute promyelocytic leukemia (APL), which is a type of blood and bone marrow cancer. It is given by I.V (intravenous, by vein). New preclinical studies have shown that when given in smaller than normal doses before treatment with chemotherapy and/or radiation therapy, the arsenic trioxide can block the activation of p53 and protect normal tissues from treatment damage. Preclinical means that the studies have been done in a laboratory and not on humans.

This study has two purposes. The first is to find the dose range for arsenic trioxide that will block p53 activity. This dose has been determined from the first five subjects who took part in the study and received arsenic trioxide. The dose of arsenic trioxide for this study is about 1/30 of the normal dose given when arsenic trioxide is used to treat acute promyelocytic leukemia. The second is to see if the arsenic trioxide will decrease the side effects of chemotherapy. In this study, arsenic trioxide is investigational. "Investigational" means that arsenic trioxide has not yet been approved by the FDA to block p53 activity.

This study will help find out what the smallest (best) dose is that can be given and the effects, good and/or bad, this drug has on people who take it. The safety of this drug in humans has been tested in prior research studies; however, whether the side effects will still be present at this lower dose is not yet known.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age with the diagnosis of malignancy other than leukemia who are to start chemotherapy known to suppress peripheral blood counts. The expected interval between each cycle of chemotherapy should be a minimum of 2 weeks. The minimum number of planned chemotherapy cycles should be 4. Radiation therapy during chemotherapy is allowed as long as less than 10% of the total bone marrow is radiated.
2. Present with or without previous treatment for the disease.
3. ECOG (Eastern Cooperative Oncology Group) performance status </= 2 (see Appendix B).
4. Life expectancy of greater than 6 months
5. Organ functions as deemed appropriate for chemotherapy per standard of care
6. Agree to use adequate contraception prior to study entry and for the duration of study participation.
7. Ability to understand and the willingness to sign a written informed consent document.
8. No baseline p53 activation in peripheral lymphocytes in culture but p53 activation should be inducible upon radiation with 2 Gy in culture

Exclusion Criteria:

1. History of allergic reactions attributed to Arsenic Trioxide
2. Experiencing uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Pregnant
4. HIV-positive patients and taking combination antiretroviral therapy.
5. History of having circulating malignant cells if the patient has lymphoma or myeloma
6. Impaired cardiac function or clinically significant cardiac diseases, including any of the following: history of long QT syndrome; mean QTc (corrected QT interval) > 500 msec on screening EKG; history of clinically manifest ischemic heart disease including myocardial infarction; stable or unstable angina, coronary arteriography or cardiac stress testing/imaging with findings consistent with coronary occlusion or infarction < 6 months prior to study start; history of heart failure or left ventricular (LV) dysfunction (LVEF < 45%) by MUGA or ECHO; clinically significant EKG abnormalities including one or more of the following: left bundle branch block (LBBB), right bundle branch block (RBBB) with left anterior hemiblock (LAHB). ST segment elevations or depressions > lmm, or 2nd (Mobitz 11) or 3rd degree AV block; history or presence of atrial fibrillation, atrial flutter or ventricular arrhythmias including ventricular tachycardia or Torsades de Pointes; other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen); clinically significant resting bradycardia (< 50 beats per minute); obligate use of a cardiac pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chul S. Ha, M.D., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Ha CS, Michalek JE, Elledge R, Kelly KR, Ganapathy S, Su H, Jenkins CA, Argiris A, Swords R, Eng TY, Karnad A, Crownover RL, Swanson GP, Goros M, Pollock BH, Yuan ZM. p53-based strategy to reduce hematological toxicity of chemotherapy: A proof of principle study. Mol Oncol. 2016 Jan;10(1):148-56. doi: 10.1016/j.molonc.2015.09.004. Epub 2015 Sep 18. PMID 26440706

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from April 2011 to November 2012. Patients were recruited from Medical Oncology clinic and due to receive standard of care chemotherapy.
Pre-assignment Details: No baseline p52 activation in peripheral lymphocytes in culture, but p53 activation inducible upon radiation in culture.
Period: Overall Study
Arm/Group | Arsenic Trioxide
Started | 50
Completed | 33
Not Completed | 17
Not completed — Withdrawal by Subject | 4
Not completed — Screen failure by p53 | 10
Not completed — Received Neulasta in one cycle | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Excluded: screen failures, withdrawals for any cause prior to completion of 2 chemotherapy cycles, or received Neulasta for only one cycle.
  Note: The 2 patients who received Neulasta for only one cycle and were not evaluable, were included in the adverse event numbers since they received study drug. Participant number will be 35 for AE module.
Arm/Group | Arsenic Trioxide
Number analyzed (Participants) | 33
Age, Continuous [Mean (Full Range); unit: years] | 52 [29 to 80]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Dose of Arsenic That Blocks Activation of p53
Description: A main objective of this trial is to find the dose of arsenic that blocks the activation of p53. Blockage will reduce the amount of p53 production as measured by Western Blot.
Time Frame: Day 1 of chemotherapy
Measure: Number; unit: mg/kg
Arm/Group | Arsenic Trioxide
Number analyzed (Participants) | 33
mg/kg | 0.005

2. Secondary Outcome: Complete Blood Count (CBC)
Description: Another objective of this trial is to assess if arsenic protects the blood counts that are adversely affected by chemotherapy
Time Frame: Day 9 of chemotherapy
Population: Data was not collected from CBC at 9 days
Groups:
- Complete Blood Count: Blood is drawn at 9 days to obtain a complete blood count
Arm/Group | Complete Blood Count
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Average time on study: 3.5 months. Reported Adverse Events (AEs) included events starting from consent to the end of final cycle of chemotherapy. Average time on study was 3.5 months with range from 2 to 6 months.
Description: If a subject experienced more than 1 of a given AE, the subject is counted only once for that AE. If a subject experienced more than one AE in a system organ class (SOC), the subject is counted only once in that SOC.
Arm/Group | Arsenic Trioxide
Serious Adverse Events (participants affected / at risk) | 9/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arsenic Trioxide (N=35)
hypotension (Vascular disorders) | 1 (1) — Not related to study drug
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to study drug
infusion site extravasation (General disorders) | 1 (1) — Not related to study drug
device related infection (Infections and infestations) | 2 (2) — Not related to study drug
non-cardiac chest pain (General disorders) | 1 (1) — Not related to study drug
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — Not related to study drug
infection, other (Infections and infestations) | 1 (1) — groin cyst, not related to study drug
lung infection (Infections and infestations) | 2 (2) — Not related to study drug
ascites (Gastrointestinal disorders) | 1 (1) — Not related to study drug
esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) — Not related to study drug
dehydration (Metabolism and nutrition disorders) | 1 (1) — Not related to study drug
sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arsenic Trioxide (N=35)
Abdominal pain (Gastrointestinal disorders) | 4
Alanine aminotransferase increased (Investigations) | 15
Alkaline phosphatase increased (Investigations) | 14
Allergic reacton (Immune system disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 22
Anemia (Blood and lymphatic system disorders) | 29
Anorexia (Metabolism and nutrition disorders) | 8
Anxiety (Psychiatric disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Aspatrate aminotransferase increased (Investigations) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 3
Blood bilirubin increased (Investigations) | 3
Blurred vision (Eye disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Breast pain (Reproductive system and breast disorders) | 2
Chills (General disorders) | 5
Constipation (Gastrointestinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Creatinine increased (Investigations) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Depression (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 7
Dizziness (Nervous system disorders) | 7
Dry mouth (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 6
Dysgeusia (Nervous system disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Ear pain (Ear and labyrinth disorders) | 2
EKG QT corrected interval prolongation (Investigations) | 14
Fatigue (General disorders) | 25
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Fever (General disorders) | 3
Flu like symptoms (General disorders) | 7
Flushing (Vascular disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, Increased appetite (Gastrointestinal disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 8
Hearing impaired (Ear and labyrinth disorders) | 2
Hot flashes (Vascular disorders) | 7
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 21
Hypocalcemia (Metabolism and nutrition disorders) | 19
Hypokalemia (Metabolism and nutrition disorders) | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 9
Hypotension (Vascular disorders) | 2
Infusion related reaction (General disorders) | 4
INR increased (Investigations) | 2
Insomnia (Psychiatric disorders) | 10
Irregular menstruation (Reproductive system and breast disorders) | 4
Lip infection (Infections and infestations) | 3
Localized edema (General disorders) | 6
Lymphocyte count decreased (Investigations) | 29
Memory impairment (Nervous system disorders) | 3
Mucosal infection (Infections and infestations) | 2
Mucositis oral (Gastrointestinal disorders) | 10
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nail discoloration (Skin and subcutaneous tissue disorders) | 8
Nail infection (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 27
Nervous System disorders-Other, Change in sense of smell (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 2
Neutrophil count decreased (Investigations) | 32
Non-cardiac chest pain (General disorders) | 2
Oral dysesthesia (Gastrointestinal disorders) | 3
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Palpitations (Cardiac disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 15
Platelet count decreased (Investigations) | 11
Pruritis (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Scalp pain (Skin and subcutaneous tissue disorders) | 6
Skin and subcutaneous tissue disorders-Other, Rash, not specified (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5
Skin infection (Skin and subcutaneous tissue disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 2
Tremor (Nervous system disorders) | 2
Upper respiratory infection (Infections and infestations) | 2
Urinary frequency (Renal and urinary disorders) | 3
Vomiting (Gastrointestinal disorders) | 7
Watering eyes (Eye disorders) | 5
Weight loss (Investigations) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
White blood cell decreased (Investigations) | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes